CLINICAL TRIAL: NCT03817580
Title: Comparative Study of Antimicrobial Effectiveness Evaluation of 26 ml Project X, 5.1 ml Project X and Prevantics® Maxi Swabstick Following ASTM E1173
Brief Title: Comparative Study of Antimicrobial Effectiveness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Professional Disposables International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ER18/282
Record Dates: First submitted 2019-01-21; First posted 2019-01-25 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Bacterial Microflora Reduction

STUDY DESIGN:
Who Masked: Participant
Masking Description: Samples are blinded to the participant and technical team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Project X 26ml (Experimental): 3.15 % w/v CHG (chlorhexidine gluconate) / 70% v/v IPA (isopropyl alcohol) contained within a saturated at use swabstick. 26ml volume. Single use.
  Interventions: Drug: Project X 26ml
- Project X 5.1ml (Experimental): 3.15 % w/v CHG (chlorhexidine gluconate) / 70% v/v IPA (isopropyl alcohol) contained within a saturated at use swabstick. 5.1ml volume. Single use.
  Interventions: Drug: Project X 5.1ml
- Prevantics Maxi Swabstick (Active Comparator): 3.15 % w/v CHG (chlorhexidine gluconate) / 70% v/v IPA (isopropyl alcohol). Swabstick. 5.1ml volume. Single use.
  Interventions: Drug: Prevantics Maxi Swabstick

INTERVENTIONS:
Drug: Project X 26ml — Application of antiseptic drug to the inguinal and abdomen areas of the subjects
  Arms: Project X 26ml
Drug: Project X 5.1ml — Application of antiseptic drug to the inguinal and abdomen areas of the subjects
  Arms: Project X 5.1ml
Drug: Prevantics Maxi Swabstick — Application of antiseptic drug to the inguinal and abdomen areas of the subjects
  Arms: Prevantics Maxi Swabstick

SUMMARY:
Comparative Study of Antimicrobial Effectiveness Evaluation of 26 ml Project X, 5.1ml Project X and Prevantics® Maxi Swabstick following ASTM E1173 - Standard Test Method for Evaluation of Preoperative, Precatheterization, or Preinjection Skin Preparations, ASTM International, West Conshohocken, PA, 2015,

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years of age and of any race
2. In good general health
3. Read, understand and sign the Informed Consent Form (ICF)
4. If female of child-bearing potential, are willing to use an acceptable method of contraception to prevent pregnancy (i.e. oral contraceptive, intra-uterine device, diaphragm, condom, abstinence, bilateral tubal ligation, or are in a monogamous relationship with a partner who has had a vasectomy)
5. Female subjects of child-bearing potential, must have a negative Urine Pregnancy Test (UPT) on Treatment Day prior to any applications of the study products
6. Screening Day Baseline microbial counts are at least 3.11 colony forming units (CFU)/cm2 bilaterally from the skin of the abdomen, and 5.00 log10 colony forming units (CFU)/cm2 bilaterally from the skin of the groin (not applicable for Neutralization study)

Exclusion Criteria:

1. Exposure of test sites to antimicrobial agents, medicated soaps, medicated shampoos, or medicated lotions, use of biocide-treated pools or hot tubs, use of tanning beds, or sunbathing during the 14-day washout conditioning period and during the test period (7-day for Neutralization study)
2. Exposure of the test sites to strong detergents, solvents, or other irritants during the 14-day washout conditioning period and during the test period (7-day for Neutralization study)
3. Wear fabric softener, bug repellent or UV-treated clothing during the 14-day washout conditioning period and during the test period (7-day for Neutralization study)
4. Receive an irritation score of 1 (any redness, swelling, rash, or dryness present at any treatment area) for any individual skin condition prior to the Screening Day baseline or Treatment Day baseline sample collection or Neutralization study
5. Use of systemic or topical antibiotic medications, steroid medications (other than for hormonal contraception or post-menopausal reasons), or any other product known to affect the normal microbial flora of the skin during the 14-day washout conditioning period and during the test period (7-day for Neutralization study)
6. Known allergies or sensitivities to vinyl, latex (rubber), alcohols, metals, inks, or tape adhesives, or to common antibacterial agents found in soaps, lotions, or ointments, particularly isopropyl alcohol or chlorhexidine gluconate
7. A medical diagnosis of a physical condition, such as a current or recent severe illness, asthma, diabetes, hepatitis, an organ transplant, mitral valve prolapses, congenital heart disease, internal prostheses, or any immunocompromised conditions such as AIDS (or HIV positive)
8. Pregnancy, plans to become pregnant within the washout and test periods of the study, or nursing a child
9. Any tattoos or scars within 2" (5.08 cm) of the test sites
10. Dermatoses, cuts, lesions, active skin rashes, or breaks or other skin disorders within 6" on or around the test sites
11. A currently active skin disease or inflammatory skin condition (for example, contact dermatitis) anywhere on the body that, in the opinion of the Consulting Physician or PI, would compromise subject safety or study integrity
12. Showering, bathing, or swimming within the 72-hour period prior to sampling for baseline screening, Treatment Day, and throughout the test period (not applicable for Neutralization study)
13. Participation in another clinical study in the past 30 days or current participation in another clinical study at time of signing informed consent
14. Any medical condition or use of any medications that, in the opinion of the PI, should preclude participation
15. Unwillingness to fulfill the performance requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rozalia Olsavszky, MD, Principal Investigator — EUROFINS EVIC PRODUCT TESTING ROMANIA S.R.L
Locations (1):
- Eurofins EVIC, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 170 individual subjects were consented, screened, treated and completed the study. Each subject is able to receive 2 test products (1 on each side of their body).
Groups:
- Project X 26ml: 3.15 % w/v CHG / 70% v/v IPA contained within a saturated at use swabstick. 26ml volume. Single use.
  Project X 26ml: Application of antiseptic drug to the inguinal and abdomen areas of the subjects
- Project X 5.1ml: 3.15 % w/v CHG / 70% v/v IPA contained within a saturated at use swabstick. 5.1ml volume. Single use.
  Project X 5.1ml: Application of antiseptic drug to the inguinal and abdomen areas of the subjects
- Prevantics Maxi Swabstick: 3.15 % w/v CHG / 70% v/v IPA. Swabstick. 5.1ml volume. Single use.
  Prevantics Maxi Swabstick: Application of antiseptic drug to the inguinal and abdomen areas of the subjects
Period: Overall Study
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick
Started | 57 | 56 | 57
Completed | 57 | 56 | 57
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick | Total
Number analyzed (Participants) | 57 | 56 | 57 | 170
Age, Continuous [Mean (Full Range); unit: years] | 58.4 [30 to 70] | 56.8 [30 to 70] | 57.6 [30 to 70] | 57.6 [30 to 70]
Sex/Gender, Customized [Number; unit: participants]
  Female | 46 | 45 | 46 | 137
  Male | 11 | 11 | 11 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 57 | 56 | 57 | 170
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Bacterial Microflora on the Inguinal Area
Description: Bacterial microflora (log10) will be measured via cup scrub method after administration of the intervention
Time Frame: 30 seconds
Population: The overall number of participants analyzed above represents the per protocol data set while the participant flow data represents the treated set. Additionally, each subject is able to receive 2 test products (1 on each side of their body).
Measure: Mean (Standard Deviation); unit: log10 CFU
Units Other Than Participants: evaluable sites
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick
Number analyzed (Participants) | 34 | 31 | 30
Number analyzed (evaluable sites) | 67 | 62 | 59
log10 CFU | -3.92 (1.42) | -3.69 (1.56) | -3.94 (1.60)

2. Primary Outcome: Change in Bacterial Microflora on the Inguinal Area
Description: Bacterial microflora (log10) will be measured via cup scrub method after administration of the intervention
Time Frame: 10 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 CFU
Units Other Than Participants: evaluable sites
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick
Number analyzed (Participants) | 34 | 31 | 30
Number analyzed (evaluable sites) | 67 | 62 | 59
log10 CFU | -4.07 (1.62) | -4.04 (1.61) | -4.17 (1.57)

3. Primary Outcome: Change in Bacterial Microflora on the Inguinal Area
Description: Bacterial microflora (log10) will be measured via cup scrub method after administration of the intervention
Time Frame: 6 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 CFU
Units Other Than Participants: evaluable sites
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick
Number analyzed (Participants) | 34 | 31 | 30
Number analyzed (evaluable sites) | 67 | 62 | 59
log10 CFU | -4.30 (1.43) | -4.57 (1.62) | -4.28 (1.53)

4. Primary Outcome: Change in Bacterial Microflora on the Abdomen
Description: Bacterial microflora (log10) will be measured via cup scrub method after administration of the intervention
Time Frame: 30 seconds
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 CFU
Units Other Than Participants: evaluable sites
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick
Number analyzed (Participants) | 30 | 30 | 32
Number analyzed (evaluable sites) | 59 | 59 | 63
log10 CFU | -3.09 (0.76) | -2.95 (1.11) | -2.85 (1.08)

5. Primary Outcome: Change in Bacterial Microflora on the Abdomen
Description: Bacterial microflora (log10) will be measured via cup scrub method after administration of the intervention
Time Frame: 10 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 CFU
Units Other Than Participants: evaluable sites
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick
Number analyzed (Participants) | 30 | 30 | 32
Number analyzed (evaluable sites) | 59 | 59 | 63
log10 CFU | -3.15 (0.85) | -2.97 (1.06) | -3.01 (0.82)

6. Primary Outcome: Change in Bacterial Microflora on the Abdomen
Description: Bacterial microflora (log10) will be measured via cup scrub method after administration of the intervention
Time Frame: 6 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 CFU
Units Other Than Participants: evaluable sites
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick
Number analyzed (Participants) | 30 | 30 | 32
Number analyzed (evaluable sites) | 59 | 59 | 63
log10 CFU | -3.19 (0.87) | -3.27 (0.95) | -3.18 (0.91)

ADVERSE EVENTS:
Time Frame: 4 months
Description: visual assessments of skin irritation and reporting of irritation by subjects
Arm/Group | Project X 26ml | Project X 5.1ml | Prevantics Maxi Swabstick
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/56 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/56 | 0/57
Other Adverse Events (participants affected / at risk) | 0/57 | 0/56 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT03817580/Prot_SAP_000.pdf